CLINICAL TRIAL: NCT04016701
Title: Immersive VR as a Tool to Support Joint Attention Skills in Children With Autism Spectrum Disorder
Brief Title: VR for Joint Attention Support in ASD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: limited recruitment within study timeline
Sponsor: Floreo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Floreo Salus Protocol 1
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Intervention (Experimental): Eight weeks of training with Floreo's VR Joint Attention Module with two sessions per week
  Interventions: Device: Floreo Joint Attention Module
- Treatment as Usual (Active Comparator): Regularly scheduled therapy
  Interventions: Behavioral: Regularly Scheduled Therapy

INTERVENTIONS:
Device: Floreo Joint Attention Module — Two sessions per week for eight weeks of the Floreo VR Joint Attention Module, delivered via a Google Cardboard compatible VR headset. Each session includes one or two 5-minute VR episodes and an intermission that is at least 3 minutes long
  Arms: VR Intervention
Behavioral: Regularly Scheduled Therapy — therapy as regularly scheduled at therapy center
  Arms: Treatment as Usual

SUMMARY:
The overall objective of this study is to determine the effectiveness of the Floreo VR Joint Attention Module in improving social communication skills in children with ASD. An additional objective is ongoing investigation of the tolerability of the product and the extent of potential adverse effects of Floreo VR, if any.

DETAILED DESCRIPTION:
The study will be a Phase II randomized controlled trial in which the Floreo VR Joint Attention Module is the intervention being evaluated. Floreo is a mobile application that offers a supervised virtual reality experience for individuals with ASD. The application provides a 3D immersive scene for Google Cardboard-compatible smartphones and a WiFi paired supervisory overview that can run on smartphones or tablets.

The therapeutic content will consist of a Learning Module focused on Joint Attention. This Joint Attention Learning Module will include separate Learning Cards (LCs) that address specific subskills necessary to develop appropriate joint attention. Each Learning Card will consist of a virtual reality environment in a safari-themed setting, complete with animals designed to draw the learner's attention when necessary.

The product will be implemented at The Children's SPOT by a therapist working with a client during the course of a therapy session.

The intervention arm participant would engage in one or two VR episodes during a scheduled session. Each episode would last no more than 5 minutes. If two episodes are done in a day, there is a mandatory break of at least 3 minutes in between them. The sessions would occur two days per week, with at least two days in between sessions to allow the eyes time to rest.

There are 15 total VR sessions in the protocol, and completion of all study sessions would take 8 weeks.

The control condition is treatment as usual, that is, regularly scheduled therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented ASD diagnosis, between 7 and 17 years of age

Exclusion Criteria:

* History of seizures, migraines, vertigo, psychosis

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Joint Attention Protocol score at 12 weeks | immediately before and 4 weeks after intervention or control period of the study
  A measure developed to rate child behaviors on 16 items involving response to joint attention and initiation of joint attention

SECONDARY OUTCOMES:
Change from Baseline Joint Attention Assessment score at 12 weeks | immediately before and 4 weeks after intervention or control period of the study
  an in-person, videotaped, play-based measure to rate frequency of joint attention skills in school-aged children. Instances of each joint attention behavior observed are summed to provide a total Joint Attention Assessment score, with higher numbers reflecting more frequent joint attention behaviors.
Change from Baseline Vineland Adaptive Behavior Scales, Third Edition total score | immediately before and 4 weeks after intervention or control period of the study
  a parent-reported measure of adaptive skills, commonly used for assessment of individuals with developmental disabilities. The Vineland provides an Adaptive Behavior Composite (ABC) score, which can be compared to a normative mean score of 100 with a normative standard deviation of 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's SPOT, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: No